CLINICAL TRIAL: NCT05777954
Title: Klotho and Bone Mineral Density (BMD) in Systemic Sclerosis Patients: Relationship with Microvascular Damage and Fibrosis
Brief Title: Klotho and Mineral Bone Density in Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mirone Luisa, Assistant Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4633
Record Dates: First submitted 2023-02-21; First posted 2023-03-21 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — two blood samples to dose DKK-1, sclerostin, Osteoprotegerin and Klotho
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Systemic Sclerosis patients: Female patients with systemic sclerosis with an age between 45 and 65 years old and did not met the exclusion criteria. Blood sample were collected to determine DKK1, Sclerostin Klotho and Osteoprotegerin. Bone mineral density was assessed. No drug was tested during the study.
  Interventions: Other: Possible Klotho effects on SSc clinical conditions, namely skeletal, fibrotic and microangiopathic damage
- Healthy subjects: Female patients with no history of inflammatory rheumatic disease and who di not met the exclusion criteria. Blood sample were collected to determine DKK1, Sclerostin Klotho and Osteoprotegerin. Bone mineral density was assessed. No drug was tested during the study.
  Interventions: Other: Evalution in healthy patients of bone mineral density, Klotho level and key bone-related cytokines

INTERVENTIONS:
Other: Possible Klotho effects on SSc clinical conditions, namely skeletal, fibrotic and microangiopathic damage — Female patients with a diagnosis of Systemic Sclerosis ( EULAR/ACR 2013 criteria ) attending the FPG Department of Rheumatology will be recruited after exclusion criteria are ruled out and informed consent is signed. DXA bone mineral density determination (Lunar Prodigy ) will be performed and bone metabolism parameters, according to routinary clinical practice, will be collected. Immunological and SSc-related disease features will also be recorded. Fibrosis will be determined by the extent of cutaneous involvement (limited or diffuse) and modified Rodnan Skin Score. Microangiopathy will be assessed by videocapillaroscopy and presence of acral ulcers or acrosteolysis; Presence of calcinosis will also be assessed .
  Upon recruitment each SSc patient will undergo blood sampling, which will be centrifuged and stored at -80° until the day of the processing. Biomarkers (Klotho, OPG, DKK, and sclerostin) will be determined using commercial kit of the ELISA Immunoenzyme techniques
  Groups: Systemic Sclerosis patients
Other: Evalution in healthy patients of bone mineral density, Klotho level and key bone-related cytokines — Healthy female control patients undergoing bone mineral density determination will be recruited upon exclusion criteria are ruled out. A detailed clinical history will be assessed and blood sempling will be processed for detection of bone-related cytokines
  Groups: Healthy subjects

SUMMARY:
The present study recruits female patients aged 45-65 years with a diagnosis of Systemic Sclerosis according to the EULAR/ACR 2013 criteria and age and gender-matched healthy control subjects. The purpose of the study is to investigate the possible role of Klotho and other cytokines involved in the osteoimmunological control of bone turnover as a possible determinant of the microvascular damage and fibrosis observed in SSc patients

DETAILED DESCRIPTION:
The present study recruits female patients aged 45-65 years with a diagnosis of Systemic Sclerosis according to the EULAR/ACR 2013 criteria and age and gender-matched healthy control subjects. The purpose of the study is to investigate the possible role of Klotho and other cytokines involved in the osteoimmunological control of bone turnover as a possible determinant of the microvascular damage and fibrosis observed in SSc patients . For each patient demographic data, history of fractures and smoking habits will be gathered. Evaluation of bone mineral density will be performed and blood samples to dose DDK1, sclerostin, osteoprotegerin and Klotho will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Systemic sclerosis diagnosis
* Signature of the informed consent

Exclusion Criteria:

* Chronic kidney disease
* Liver or thyroid disease
* Diabetes
* Ongoing diuretic treatment
* Estrogen replacing treatment
* Vitamin D or Calcium supplementation
* Drugs able to interfere with bone turn-over (such as bisphosphonates or glucocorticoids)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with a diagnosis of Systemic Sclerosis according to the EULAR/ACR 2013 criteria and followed by the FPG-IRCSS Rheumatology Department will be progressively recruited, after exclusion criteria are ruled out and informed consent is signed.
  Concomitantly healthy control female patients undergoing bone mineral density determination are recruited, once exclusion criteria are ruled out.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Klotho serum levels in a group of 63 female SSc patients aged 45-65 years compared to 63 age and sex-matched healthy controls | 21 months
  Klotho serum levels in each SSc and control subject will be determined by a commercial ELISA assay

SECONDARY OUTCOMES:
Klotho serum levels in female SSc patients: relationship to microvascular damage and fibrosis | 21 months
  Evaluation of a possible relationship among Klotho serum levels, the extent and type of the microvascular damage assessed by videocapillaroscopy, and the extent of the cutaneous fibrotic involvement assessed by the modified Rodnan skin score (mRSS).
Klotho serum levels in female SSc patients: relationship to bone mineral density values | 21 months
  Detection of a possible relationship between Klotho serum levels and bone mineral density values in female SSc patients stratified according to the extent of vascular and fibrotic damage
Klotho serum levels in female SSc patients relationship to key bone-related cytokine serum levels | 21 months
  Assessment of a possible relationship among Klotho, DDK-1, OPG, and sclerostin serum levels

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Mirone, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Division of Rheumatology, Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No